CLINICAL TRIAL: NCT00273650
Title: Double-Blind Placebo Controlled, Cross-over Trial of Subcutaneous B12 on Behavioral and Metabolic Measures in Children With Autism.
Brief Title: Efficacy Study of Subcutaneous Methyl-B12 in Children With Autism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MB12-AUT
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Autistic Disorder
Keywords: Autism; Placebo; B12; Controlled; Complementary Alternative Medicine; Vitamin Supplement
MeSH Terms: conditions — Autistic Disorder | interventions — mecobalamin; Vitamin B 12; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Methyl-B12
  Interventions: Drug: methylcobalamin
- B (Placebo Comparator): Saline placebo
  Interventions: Other: saline placebo

INTERVENTIONS:
Drug: methylcobalamin — Methylcobalamin (25,000μg/ml), at a dosage of 64.5μg/kg, or saline placebo administered subcutaneously, once every three days for six weeks. At six weeks, subjects cross over to the other treatment given every three days for another six weeks. Post 12 weeks, treatment with open label methylcobalamin will continue once every three days, for six months.
  Other Names: Vitamin B-12; Methyl-B12
  Arms: A
Other: saline placebo — Methylcobalamin (25,000μg/ml), at a dosage of 64.5μg/kg, or saline placebo administered subcutaneously, once every three days for six weeks. At six weeks, subjects cross over to the other treatment given every three days for another six weeks. Post 12 weeks, treatment with open label methylcobalamin will continue once every three days, for six months.
  Other Names: saline
  Arms: B

SUMMARY:
We will be testing a specific dietary supplement, methylcobalamin (vitamin B12). Follow-up assessments with our clinical team will take place over the 12-week study period so that we can record any changes in development. The main goal of this study is to determine if subcutaneous injections of vitamin B12 given every three days can positively affect behavior and development in children with autism.

Hypothesis: Methylcobalamin injections will improve measures of executive function, speech, and socialization in children with autism, and will be associated with metabolic improvement.

DETAILED DESCRIPTION:
Autism is a complex neurodevelopmental disorder that is thought to involve an interaction between multiple and variable susceptibility genes (Keller & Persico, 2003), epigenetic effects (Beaudet, 2002), and environmental factors (London, 2000). The increase in the prevalence of autistic spectrum disorders from 4-5/10,000 in the 1980s to 30-60/10,000 in the last decade has raised great concern (Bertrand et al., 2001; DeStefano et al., 2004; Steinhausen et al., 1986; Yeargin-Allsopp et al., 2003). Research into potential therapeutic interventions designed to ameliorate the metabolic and clinical symptoms of autism is urgently needed to reduce the enormous public health burden of this disorder and to improve the quality of life for affected children and their families. Nutritional supplementation through subcutaneous injections of methyl B12 is a current treatment for children with autism that has anecdotal reports of remarkable clinical improvements and few side effects. However there are no published studies to support its clinical benefit.

Comparison: Injections of methylcobalamin compared to injections of sterile saline over a six week period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DSM IV defined autism and meets cut off on Autism Diagnostic Inventory-Revised (ADI-R) and the Autism Diagnostic Observation Scale (ADOS).
* Age 3 to 8 years
* IQ of 50 or above
* Willingness of parents to administer subcutaneous methyl B12.
* Parental agreement to continue present dietary, behavioral or psychotropic drug treatment but not change treatment during 12 week intervention or wait list.

Exclusion Criteria:

* Clinical evidence of seizure disorder
* Cancer
* Recent surgery
* Active infection with fever
* Fragile X or other known genetic cause of autism
* Bleeding disorder
* Perinatal brain injury (e.g. cerebral palsy)
* Current use of any methyl B12 product
* Evidence for malnutrition seen in abnormal albumin level

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2005-07; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Primary measure is the Clinical Global Impression Scale -Improvement supplemented by videos taken at all visits and rated blindly to measure executive function, speech, and language, and socio-economic development. | 12 Weeks to 6 Months

SECONDARY OUTCOMES:
Secondary measures:NEPSY, ABC, PPVT, SB:V, PDRF, MCDI, PIA-CV, and CARS. | 12 Weeks to 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Hendren, D.O., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaudet AL. Is medical genetics neglecting epigenetics? Genet Med. 2002 Sep-Oct;4(5):399-402. doi: 10.1097/00125817-200209000-00013. No abstract available. PMID 12394355
- [Background] Bertrand J, Mars A, Boyle C, Bove F, Yeargin-Allsopp M, Decoufle P. Prevalence of autism in a United States population: the Brick Township, New Jersey, investigation. Pediatrics. 2001 Nov;108(5):1155-61. doi: 10.1542/peds.108.5.1155. PMID 11694696
- [Background] DeStefano F, Bhasin TK, Thompson WW, Yeargin-Allsopp M, Boyle C. Age at first measles-mumps-rubella vaccination in children with autism and school-matched control subjects: a population-based study in metropolitan atlanta. Pediatrics. 2004 Feb;113(2):259-66. doi: 10.1542/peds.113.2.259. PMID 14754936
- [Background] Esch BE, Carr JE. Secretin as a treatment for autism: a review of the evidence. J Autism Dev Disord. 2004 Oct;34(5):543-56. doi: 10.1007/s10803-004-2549-6. PMID 15628608
- [Background] Finkelstein JD. Pathways and regulation of homocysteine metabolism in mammals. Semin Thromb Hemost. 2000;26(3):219-25. doi: 10.1055/s-2000-8466. PMID 11011839
- [Background] Gulati S, Brody LC, Banerjee R. Posttranscriptional regulation of mammalian methionine synthase by B12. Biochem Biophys Res Commun. 1999 Jun 7;259(2):436-42. doi: 10.1006/bbrc.1999.0696. PMID 10362526
- [Background] Keller F, Persico AM. The neurobiological context of autism. Mol Neurobiol. 2003 Aug;28(1):1-22. doi: 10.1385/MN:28:1:1. PMID 14514983
- [Background] Levy SE, Mandell DS, Merhar S, Ittenbach RF, Pinto-Martin JA. Use of complementary and alternative medicine among children recently diagnosed with autistic spectrum disorder. J Dev Behav Pediatr. 2003 Dec;24(6):418-23. doi: 10.1097/00004703-200312000-00003. PMID 14671475
- [Background] London EA. The environment as an etiologic factor in autism: a new direction for research. Environ Health Perspect. 2000 Jun;108 Suppl 3(Suppl 3):401-4. doi: 10.1289/ehp.00108s3401. PMID 10852835
- [Background] Miller AL. The methionine-homocysteine cycle and its effects on cognitive diseases. Altern Med Rev. 2003 Feb;8(1):7-19. PMID 12611557
- [Background] Muntjewerff JW, van der Put N, Eskes T, Ellenbroek B, Steegers E, Blom H, Zitman F. Homocysteine metabolism and B-vitamins in schizophrenic patients: low plasma folate as a possible independent risk factor for schizophrenia. Psychiatry Res. 2003 Nov 1;121(1):1-9. doi: 10.1016/s0165-1781(03)00200-2. PMID 14572619
- [Background] Pogribna M, Melnyk S, Pogribny I, Chango A, Yi P, James SJ. Homocysteine metabolism in children with Down syndrome: in vitro modulation. Am J Hum Genet. 2001 Jul;69(1):88-95. doi: 10.1086/321262. Epub 2001 Jun 5. PMID 11391481
- [Background] Schulz JB, Lindenau J, Seyfried J, Dichgans J. Glutathione, oxidative stress and neurodegeneration. Eur J Biochem. 2000 Aug;267(16):4904-11. doi: 10.1046/j.1432-1327.2000.01595.x. PMID 10931172
- [Background] Sogut S, Zoroglu SS, Ozyurt H, Yilmaz HR, Ozugurlu F, Sivasli E, Yetkin O, Yanik M, Tutkun H, Savas HA, Tarakcioglu M, Akyol O. Changes in nitric oxide levels and antioxidant enzyme activities may have a role in the pathophysiological mechanisms involved in autism. Clin Chim Acta. 2003 May;331(1-2):111-7. doi: 10.1016/s0009-8981(03)00119-0. PMID 12691871
- [Background] Steinhausen HC, Gobel D, Breinlinger M, Wohlleben B. A community survey of infantile autism. J Am Acad Child Psychiatry. 1986 Mar;25(2):186-9. doi: 10.1016/s0002-7138(09)60225-9. No abstract available. PMID 3486202
- [Background] Sturmey P. Secretin is an ineffective treatment for pervasive developmental disabilities: a review of 15 double-blind randomized controlled trials. Res Dev Disabil. 2005 Jan-Feb;26(1):87-97. doi: 10.1016/j.ridd.2004.09.002. PMID 15590241
- [Background] Yeargin-Allsopp M, Rice C, Karapurkar T, Doernberg N, Boyle C, Murphy C. Prevalence of autism in a US metropolitan area. JAMA. 2003 Jan 1;289(1):49-55. doi: 10.1001/jama.289.1.49. PMID 12503976
- [Background] Yorbik O, Sayal A, Akay C, Akbiyik DI, Sohmen T. Investigation of antioxidant enzymes in children with autistic disorder. Prostaglandins Leukot Essent Fatty Acids. 2002 Nov;67(5):341-3. doi: 10.1054/plef.2002.0439. PMID 12445495